CLINICAL TRIAL: NCT04394702
Title: Efficacy of One-Shape Single-file System in Pulpectomy of Infected Primary Molars: In-vitro and In-vivo Randomized Controlled Trial.
Brief Title: Single-file Pulpectomy in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Osama Seif El-Nasr Hussein Gad El-Hak, assistant lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 42/183/11/2016
Record Dates: First submitted 2020-05-10; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Pulpal Necrosis
Keywords: Pulpectomy; Pediatric Dentistry
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One Shape Single-file rotary system (Experimental)
  Interventions: Other: One Shape Single-file rotary system
- Manual stainless steel K-file (Active Comparator)
  Interventions: Other: manual stainless steel K-file

INTERVENTIONS:
Other: One Shape Single-file rotary system — rotational single file system used for mechanical debridement of root canals
  Arms: One Shape Single-file rotary system
Other: manual stainless steel K-file — sequential manual filing with stainless steel K-files
  Arms: Manual stainless steel K-file

SUMMARY:
The current study evaluates the rotational One Shape single-file system regarding clinical and radiographic outcomes in root canal treatment of infected primary molars.

This randomized clinical trial was carried out on 94 primary molars on children in the age group from 4 to 6 years. The teeth selected for this study were randomly assigned into 2 groups according to the used endodontic preparation system. Group I: 47 primary molars were instrumented with One Shape rotational single-file system. Group II: 47 primary molars were instrumented with stainless steel K-files. All teeth were evaluated clinically and radigraphically for 12 months with periodic recall at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Children categorized as class I or II according to American Society of Anesthesiologists (ASA).
* Children aged between 4 and 6 years with at least one necrotic primary second mandibular molar.
* History of dull toothache over an extended period of time
* History of spontaneous pain or pain at night
* Swelling adjacent to tooth with or without a sinus tract
* Abnormal tooth mobility
* Presence of necrotic pulp tissue or purulent discharge when the pulp chamber was accessed
* Interruption of lamina dura or thickening of periodontal ligament space
* Furcational radiolucency did not surpass half of the distance between the furcation and permanent successor
* Negative findings of internal root resorption
* External root resorption confined to the apical third and with at least two-thirds of the root length was intact

Exclusion Criteria:

* Uncoperative children or parents/legal guardians
* Sever intellectual, behaviour or emotional problems
* Non-restorable tooth crowns
* Root canal obliteration
* Presence of underlying dentigerous or follicular cysts

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Pain presence or absence | one year
  score 0 was applied for absence of pain and score 1 was applied for presence of pain
swelling presence or absence | one year
  score 0 was applied for absence of swelling and score 1 was applied for presence of swelling
radiographic success or failure | one year
  it was done using periapical radiograph and score 0 was applied for absence of radiolucency and score 1 was applied for presence of radiolucency

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Faculty of Dentistry., Minya, Egypt